CLINICAL TRIAL: NCT02444455
Title: Safety and Efficacy of Human Umbilical-Cord-Derived Mesenchymal Stem Cell Transplantation in Acute Lung Injury
Brief Title: Human Umbilical-Cord-Derived Mesenchymal Stem Cell Therapy in Acute Lung Injury
Acronym: UCMSC-ALI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Ivy Institute of Stem Cells Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-IVY-SC-003
Record Dates: First submitted 2015-05-08; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: cellular therapy; acute lung injury; acute respiratory distress snydrome; human umbilical cord mesenchymal stem cell; phase 1/2 clinical study; allogeneic stem cell transplantation; ALI; ARDS
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UCMSC group (Experimental): Human umbilical cord MSCs are administrated to patients by intravenous infusion
  Interventions: Biological: UCMSC group

INTERVENTIONS:
Biological: UCMSC group — Human umbilical cord MSCs are transplanted by intravenous infusion(5×10^5/kg) once a day,a total of three times.

SUMMARY:
Phase I-II Clinical Trial - Safety and efficacy of umbilical-cord-derived mesenchymal stem cell (UC-MSC) in patients with Acute Lung Injury ,open label, controlled prospective study.

DETAILED DESCRIPTION:
Phase I-II Clinical Trial - Safety and efficacy of umbilical-cord-derived mesenchymal stem cell (UC-MSC) in patients with acute lung injury,open label, controlled prospective study.

Every patient will maintain their standard treatment of acute lung injury, with maximum tolerated dosage without side effects.

The day of infusion will be considered day zero. From that moment, followup will be divided into 2,7,14 days.

Clinical results will be analyzed after completion of 14 days of followup.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 35 and 70 y
* Acute onset within 7 days.
* Oxygenation index:200<PaO2/FiO2≤300mmHg; alveolar-arterial oxygen differences:P(A-a)O2>35mmHg
* Bilateral infiltrates on chest radiography
* No cardiac failure

Exclusion Criteria:

* Declined to sign informed consent
* Socially and mentally disabilities
* Malignant diseases
* Combined with severe infectious diseases
* Patients with positive blood tests for Hepatitis B or Hepatitis C or HIV or tuberculosis at the time of screening
* Pregnant or perinatal women
* Severe diseases of any major organs

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety will be determined by the assessment of major adverse events | From day 0 at the start of treatment to day 14.
  Safety will be determined by the assessment of major adverse events defined as death, and the incidence of prespecified infusion-associated events and non-serious adverse events thought to be related to the MSC infusion.

SECONDARY OUTCOMES:
Quantify pulmonary respiratory function measured by chest computerized tomography | Participants will be followed for the duration of hospital,2 day post-infusion, and days 7,14.
The efficacy of UC-MSC treatment was measured by arterial blood gas analysis | Participants will be followed for the duration of hospital,2 day post-infusion, and days 7,14.
The efficacy of UC-MSC treatment was measured by biological markers,including markers of inflammation，IL-6 | 6 hours post-infusion, and days 1, 2, and 3
The efficacy of UC-MSC treatment was measured by biological markers,including markers of inflammation，IL-8 | 6 hours post-infusion, and days 1, 2, and 3

CONTACTS AND LOCATIONS:
Overall Officials: Bing Liu, M.D., Study Chair — 307-IVY Translational Medicine Center; Changqing Bai, M.D., Study Director — Department of Respiration, Affiliated Hospital to Academy of Military Medical Sciences; Huiying Liu, M.D., Principal Investigator — Department of Respiration, Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of Respiration,Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China